CLINICAL TRIAL: NCT03267446
Title: The Role of Grey Scale Ultrasound, 2D, and 3D Power Doppler in Diagnosing and Predicting the Surgical Risks in Patients With Morbidly Adherent Placenta.
Brief Title: Doppler Imaging and Morbidly Adherent Placenta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Hussein, Assistant Professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CU28817
Record Dates: First submitted 2017-08-29; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Antepartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional group (Experimental): Patients confirmed having one or more of the signs of morbidly adherent placenta will be examined by 3D Ultrasound and 3D power Doppler. Patients will then be prepared for the operation.Cesarean hysterectomy will be done with removal of the uterus and the placenta as one mass.Cases with focal invasion of the uterus will be given a trial for conservative management. The whole specimen will be sent for histopathological examination, and the determination of length and depth of invasion.
  Interventions: Device: 3D Doppler Ultrasound

INTERVENTIONS:
Device: 3D Doppler Ultrasound — 3D volumes will be obtained in automatic sweeps using a motorized curved-array transducer while the women held their breath. In order to interpret the data consistently, the settings of power, On Voluson E10; GE Medical Systems)

SUMMARY:
The aim of this study is to assess the value of adding 3D power Doppler (as a diagnostic technique) to gray scale technique in the antenatal diagnosis of morbidly adherent placenta as well as predict the surgical outcome regarding the type of surgery and the intra operative morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 45.
* Pregnant 32 weeks or more.
* Placenta previa (Major and Minor).
* History of previous cesarean section.

Exclusion Criteria:

* Medical disorders such as bleeding disorders.
* Lethal fetal anomalies.
* Delivery before 34 weeks.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of 3D power Doppler in detecting morbidly adherent placenta. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Hussein, MD, Principal Investigator — Cairo Univeristy
Locations (1):
- Kasr el aini hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided